CLINICAL TRIAL: NCT04826536
Title: Treatment Patterns and Outcomes Study for Psoriasis (PSO) in Japan
Brief Title: A Study of Treatment Patterns and Clinical Outcomes of Psoriasis in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-166
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
Keywords: Japan; Observational; Psoriasis; Retrospective
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with psoriasis

SUMMARY:
The purpose of this study is to understand current real-world treatment patterns and clinical outcomes, reasons for switching treatment, and participant characteristics using each systemic psoriasis treatment in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriasis
* Can be followed for at least 2 years
* Treated with any of the following systemic therapy for psoriasis at time of follow-up start: Tumor Necrosis Factor (TNF) inhibitors (infliximab, adalimumab, and certolizumab pegol), Interleukin (IL)-12/23 inhibitors (ustekinumab), IL-23 inhibitors(guselkumab, risankizumab, and tildrakizumab), IL-17 inhibitors (secukinumab, ixekizumab, and brodalumab), Apremilast, Methotrexate, Cyclosporine, Etretinate

Exclusion Criteria:

* Enrolled in any clinical trials for psoriasis in their follow-up period
* Developed psoriatic arthritis, guttate psoriasis, erythrodermic psoriasis, and pustular psoriasis at time of start date
* Treated with any of the following systemic therapy before they were diagnosed with psoriasis: TNF inhibitors (infliximab, adalimumab, and certolizumab pegol), IL-12/23 inhibitors (ustekinumab), IL-23 inhibitors(guselkumab, risankizumab, and tildrakizumab), IL-17 inhibitors (secukinumab, ixekizumab, and brodalumab), Apremilast, Methotrexate, Cyclosporine, Etretinate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 participants, from 2 to 4 institutes which have a central role of psoriasis therapy in Japan, will be entered into the study if they started systemic treatment after 01/01/2017 and followed until either 12/31/2020, death, or lost to follow-up, whichever occurs first.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Distribution of participant background at first visit: Age | At Baseline
Distribution of participant background at first visit: Sex | At Baseline
Distribution of participant background at first visit: Duration with psoriasis | At Baseline
Distribution of participant background at first visit: Comorbidities | At Baseline
Distribution of participant background at first visit: Current status of phototherapy | At Baseline
Treatment patterns: Drug names treated during study period | Up to 4 years
Treatment patterns: Drug categories treated during study period | Up to 4 years
Treatment patterns: Number of treatment changes during study period | Up to 4 years
Treatment patterns: Treatment duration of each drug during study period | Up to 4 years
Treatment patterns: Duration between withdrawal of one drug and start of a new drug during study period | Up to 4 years
Treatment patterns: Adverse event (AE) at time of withdrawal of some drug | Up to 4 years
Treatment patterns: Psoriasis area severity index (PASI) at time of withdrawal | Up to 4 years
Treatment patterns: PASI at time of start of a new drug | Up to 4 years
Treatment patterns: PASI improvement from start of one drug to withdrawal of other drug | Up to 4 years
Treatment patterns: Reason for treatment change during study period | Up to 4 years
Treatment patterns: Status of phototherapy combination with systemic treatment | Up to 4 years

SECONDARY OUTCOMES:
Distribution of comorbidities that affect treatment choice and change | Up to 4 years
Distribution of AEs that affect treatment choice and change | Up to 4 years
Mean number of drug changes until participants achieve PASI 75 during study period | Up to 4 years
  75% reduction in the Psoriasis Area and Severity Index score (PASI 75)
Mean number of drug changes until participants achieve PASI 90 during study period | Up to 4 years
  90% reduction in the Psoriasis Area and Severity Index score (PASI 90)
Mean number of drug changes until participants achieve PASI 100 during study period | Up to 4 years
  100% reduction in the Psoriasis Area and Severity Index score (PASI 100)
Total period until participants achieve PASI 75 during study period | Up to 4 years
Total period until participants achieve PASI 90 during study period | Up to 4 years
Total period until participants achieve PASI 100 during study period | Up to 4 years
Mean period of participants achieve PASI 75 by each systemic treatment | Up to 4 years
Mean period of participants achieve PASI 90 by each systemic treatment | Up to 4 years
Mean period of participants achieve PASI 100 by each systemic treatment | Up to 4 years
Description of relationship between the reasons for treatment change and period of withdrawal | Up to 4 years
Efficacy after re-start treatment measured by PASI | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm